CLINICAL TRIAL: NCT03987711
Title: Strategies for the Management of Atrial Fibrillation in patiEnts Receiving Dialysis (SAFE-D)
Brief Title: Strategies for the Management of Atrial Fibrillation in patiEnts Receiving Dialysis
Acronym: SAFE-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The George Institute for Global Health (Sydney, Australia) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAFE-D-01
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation; End Stage Renal Failure on Dialysis
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Warfarin (Experimental): Individuals randomized to this arm will be exposed to dose-adjusted daily warfarin targeting an international normalized ratio (INR) of 2.0-3.0.
  Interventions: Drug: Warfarin
- Apixaban (Active Comparator): Individuals randomized to this arm will receive apixaban 5 mg twice daily (a reduced dose of 2.5 mg twice daily will be given to selected participants).
  Interventions: Drug: Apixaban
- No oral anticoagulation (Active Comparator): Individuals in this arm will be exposed to a treatment strategy in which no oral anticoagulation is prescribed.
  Interventions: Other: No oral anticoagulation

INTERVENTIONS:
Drug: Warfarin — Individuals randomized to this arm will be exposed to dose-adjusted daily warfarin targeting an international normalized ratio (INR) of 2.0-3.0.
  Other Names: Coumadin
  Arms: Warfarin
Drug: Apixaban — Individuals randomized to this arm will receive apixaban 5 mg twice daily (a reduced dose of 2.5 mg twice daily will be given to selected participants).
  Other Names: Eliquis
  Arms: Apixaban
Other: No oral anticoagulation — No oral anticoagulation
  Arms: No oral anticoagulation

SUMMARY:
The prevention of atrial fibrillation related thromboembolism in the dialysis population is unclear. While the practice of anticoagulation appears favorable in patients with mild-to-moderate chronic kidney disease, no patients with severe chronic kidney disease (estimated glomerular filtration rate <25 ml/min), and specifically those receiving dialysis, have been included in randomized trials.Moreover, the effect of anticoagulation in the dialysis population may fundamentally differ from those studied in clinical trials. Accordingly, characterization of the optimal management strategy to reduce the risk of stroke and systemic embolism in patients with atrial fibrillation receiving dialysis is a priority. The overall goal of this pilot trial is to evaluate the feasibility of conducting a randomized controlled trial comparing anticoagulation strategies in patients with atrial fibrillation receiving dialysis (either hemodialysis or peritoneal dialysis).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Receiving maintenance hemodialysis or peritoneal dialysis for > 90 days.
3. History of AF or atrial flutter as defined by:

   (i) AF or atrial flutter on a 12 lead ECG at enrollment, and not due to a reversible cause, or (ii) AF or atrial flutter documented on two separate occasions, not due to a reversible cause, at least 1 day apart prior to enrollment. AF or atrial flutter may be documented by ECG, or as an episode lasting at least 30 seconds on a rhythm strip or Holter recording, or more than 30 minutes if using pacemaker or implantable cardioverter defibrillator (ICD) recordings, or (iii) AF or atrial flutter documented on one occasion, not due to a reversible cause, prior to enrollment and being treated with an oral anticoagulant for AF or atrial flutter at enrollment. [AF or atrial flutter may be documented by ECG, or as an episode lasting at least 30 seconds on a rhythm strip or Holter recording, or more than 30 minutes if using pacemaker or implantable cardioverter defibrillator (ICD) recordings, or mentioned in the medical record], or (iv) AF or atrial flutter documented on one occasion on ECG, not due to a reversible cause, prior to enrollment and at least one more episode of AF or atrial flutter mentioned in the medical record, or (v) AF or atrial flutter documented on one occasion in a cardiologist report, not due to a reversible condition, prior to enrollment.
4. Satisfying CHADS-65 criteria: i) Age ≥65 or ii) Age <65 and one of: hypertension, diabetes mellitus, congestive heart failure, stroke/transient ischemic attack or peripheral embolism.

Exclusion Criteria:

1. Moderate or severe mitral stenosis.
2. Conditions other than non-valvular atrial fibrillation that require oral anticoagulation, such as mechanical prosthetic valve, deep venous thrombosis, or pulmonary embolism.
3. Need for aspirin at a dose > 165 mg a day, or need for aspirin in combination with P2Y12 antagonist therapy.
4. Need for an interacting drug which precludes the safe use of apixaban.
5. Life expectancy < 6 months.
6. Scheduled live-donor kidney transplant in the next 6 months.
7. A woman who is pregnant or breastfeeding or unwilling to pursue methods of contraception if < 12 months since the last menstrual period.
8. Co-enrollment in a clinical trial where the intervention is deemed to interfere with the adherence, safety or efficacy of the intervention provided herein.
9. Patient's attending physician(s) (e.g., nephrologist and/or cardiologist and/or neurologist) believes that oral anticoagulation is absolutely mandated.
10. Patient's attending physician(s) (e.g., nephrologist and/or cardiologist and/or neurologist) believes that oral anticoagulation is absolutely contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment of the target population within 2 years | 2 years from start of trial
At least 80% of randomized participants remain in the trial and on the allocated study treatment at the end of the 26-week study period. | 26 weeks

SECONDARY OUTCOMES:
Proportion of patients randomized to warfarin achieving a Time in the Therapeutic Range (TTR) >65%. | 26 weeks
>95% of randomized patients adhere to the enrollment criteria with respect to atrial fibrillation or atrial flutter | End of trial
  Through adjudication of ECGs or other cardiac diagnostics
Major bleeding | 26 weeks
  As defined by the International Society of Thrombosis and Haemostasis (ISTH)
Clinically relevant non-major bleeding | 26 weeks
  As defined by the International Society of Thrombosis and Haemostasis (ISTH)
Stroke and systemic embolism | 26 weeks
All cause mortality | 26 weeks
Non-fatal myocardial infarction | 26 weeks
Vascular events not related to dialysis access | 26 weeks
Events of special interest related to dialysis access, the dialysis procedure or the oral anticoagulants | 26 weeks
  Thrombosis of fistula or graft; fistula or graft abandonment; thrombosis of dialysis catheter; red blood cell transfusions; calciphylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Ziv Harel, Principal Investigator — Unity Health Toronto; Ron Wald, Principal Investigator — Unity Health Toronto
Locations (28):
- Australia (4):
  - Nepean Hospital, Kingswood, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - St. George Hospital, Sydney
- Canada (24):
  - Surrey Memorial Hospital, Surrey, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Seven Oaks General Hospital, Winnipeg, Manitoba
  - Nova Scotia Health Authority, QEII Health Sciences Centre, Halifax, Nova Scotia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Halton Healthcare - Oakville Trafalgar Memorial Hospital, Oakville, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - The Ottawa Hospital - Riverside Campus, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health Toronto, at its St. Michael's Hospital site, Toronto, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - St. Joseph's Health Centre Toronto, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec, Quebec
  - Regina General Hospital, Regina, Saskatchewan

REFERENCES:
- [Derived] Harel Z, Smyth B, Badve SV, Blum D, Beaubien-Souligny W, Silver SA, Clark E, Suri R, Mavrakanas TA, Sasal J, Prasad B, Eikelboom J, Tennankore K, Rigatto C, Prce I, Madore F, Mac-Way F, Steele A, Zeng Y, Sholzberg M, Dorian P, Yan AT, Sood MM, Gladstone DJ, Tseng E, Kitchlu A, Walsh M, Sapir D, Oliver MJ, Krishnan M, Kiaii M, Wong N, Kotwal S, Battistella M, Acedillo R, Lok C, Weir M, Wald R. Anticoagulation for Patients with Atrial Fibrillation Receiving Dialysis: A Pilot Randomized Controlled Trial. J Am Soc Nephrol. 2025 May 1;36(5):901-910. doi: 10.1681/ASN.0000000000000495. Epub 2024 Nov 4. PMID 39495569